CLINICAL TRIAL: NCT04321629
Title: Autologous Adipose Tissue Injection Versus Platelet-rich Plasma (PRP) Injection in the Treatment of Knee Osteoarthritis: a Randomized, Controlled Study - Study Protocol
Brief Title: Knee Arthritis Treatment With Autologous Fragmented Adipose Tissue and PRP - Comparison of Two Treatment Methods
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rehasport Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSC_PBAK_2018_V3
Record Dates: First submitted 2020-03-20; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Osteo Arthritis Knee; Knee Osteoarthritis; Knee Pain Chronic; Knee Arthritis; Knee Disease; Knee Pain Swelling; Joint Diseases
Keywords: knee; arthritis; prp; msc; fat transfer; adipose tissue
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases; Arthritis; Insomnia, Fatal Familial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous Fat Tissue Group (Experimental): Group of patients treated with intra-articular injections of autologous adipose tissue.
  Interventions: Combination Product: autologous adipose tissue transfer
- PRP Group (Active Comparator): Group of patients treated with intra-articular injections of platelet-rich-plasma.
  Interventions: Combination Product: PRP injections

INTERVENTIONS:
Combination Product: autologous adipose tissue transfer — experimental group: liposuction, adipose tissue preparation and intra-articular injection
  Arms: Autologous Fat Tissue Group
Combination Product: PRP injections — control group: blood collection, blood preparation and intra-articular PRP injection
  Arms: PRP Group

SUMMARY:
This is a prospective, randomized, controlled study. The purpose of this study is to assess functional and clinical changes among patients with symptomatic knee OA treated with intra-articular injections of autologous adipose tissue or PRP and to compare the efficacy of both therapeutic methods. We hypothesize that adipose tissue injections will improve patients' quality of life and functional status and will decrease pain level significantly more than PRP injections. In addition to the functional tests and muscle strength measurement, the patient reported outcome measures (PROMs) of the knee joint function and quality of life will be used to assess each participant.

The same inclusion criteria have been established for an Experimental Group (subjects treated with autologous fat tissue) and a Control Group (subjects treated with PRP). Those criteria consist of: symptomatic knee OA, age between 45 and 65 y.o., Kellgren- Lawrence grades I - III OA, no or minimal positive effects of previous conservative treatment (rehabilitation, hyaluronic acid injections, steroid injections). Those patients who meet inclusion criteria will be allocated to Fat Tissue Group or PRP Group randomly.

Patients will be assessed five times: before treatment and 1, 3, 6 and 12 months after the treatment. The PROMs consist of the four questionnaires: The Knee injury and Osteoarthritis Outcome Score (KOOS), International Knee Documentation Committee 2000 (IKDC 2000), the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) (21,22), the Health Questionnaire EQ- 5D- 5L.

Moreover, three functional tests will be performed to assess patient's functional status: The Timed Up and Go Test (TUG), The 5 Times Sit to Stand Test (5xSTS), The 10m Walk Test (10mWT). To assess strength parameters of the knee flexors and extensors the Maximal Voluntary Isometric Contraction (MVIC) will be measured. Each test will be supervised by the same one physiotherapist to avoid any interexaminer bias and discrepancies during testing.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled study. The purpose of this study is to assess functional and clinical changes among patients with symptomatic knee OA treated with intra-articular injections of autologous adipose tissue or PRP and to compare the efficacy of both therapeutic methods.

Lipoaspiration procedure Lipoaspiration will take place in the operating room under general anesthesia for patient's and doctor's comfort. The most frequent donor site is abdomen (14,15). The patient will be placed in a supine position. At first, two small incisions at the level of umbilicus will be made by the trained orthopaedic surgeon (TP or PB). Then Klein solution (saline with lidocaine and epinephrine) will be infused to reduce bleeding. Ten minutes is required for infiltration. Next step is a liposuction performed with a thin cannula inserted through incisions. Finally, skin sutures and the pressure dressing will be applied. To minimize risk of bleeding and hematoma, an elastic belt will be recommended, as well as partial weight bearing within first two weeks. Harvested adipose tissue will be prepared in a Lipogems kit (14). The final product will be transferred into 10-ml syringes. About 10 ml of the product will be injected into the affected knee joint.

PRP procedure PRP preparation takes place in an outpatient clinic. 10-ml sterile collecting tubes containing citrate will be placed in a centrifuge (Centrifuge MPV- 223e) with a tilting rotor. Rotation will last 7 minutes at 2054 rounds per minute. After centrifugation, PRP will be collected up to 3 ml for separate 10-ml syringe. 3 ml of PRP will be injected into the knee joint. Procedure will be repeated three times in 7 day interval.

Injection procedure Joint injection will be performed by TP or PB in the same manner for both groups: patient placed in supine position, affected knee extended, a 21-Gauge needle inserted into the suprapatellar pouch, in case of joint effusion - aspiration of synovial fluid and finally administration of autologous fat tissue or PRP.

This study protocol has several strengths and weaknesses. Undoubtedly one of strongest point of this study is wide, multidimensional functional assessment, which will give a large amount of objective data. To our knowledge, this research is the first one which includes the battery of functional tests and MVIC as an outcome measurement tool. This study will use 4 questionnaires, including WOMAC, which is described by physicians as a gold standard for assessing the effectiveness of knee OA treatment (47,48).

On the other hand this study has several limitations. Primarily - the lack of blinding and we consider this as a risk of both, subject and investigator bias. Next and equally important limitation is a small size of the study. Furthermore, autologous fat tissue procedure is definitely more invasive and more stressful for the patients than PRP procedure. Hence, taking all into consideration, to adopt autologous fat tissue as a knee OA therapy, based on the future results, we have to detect definite, statistically significant and clinically noticeable difference.

Our PRP procedure gives us the possibility to examine the patient and assess the reaction to intra- articular injection 3 times (3 injections) in 7 day interval. These visits are often associated with physical therapy, which consists of manual therapy and individualized exercise program. Autologous fat tissue procedure does not give us such a possibility. The doctor and physiotherapist see the patient on the day of the surgery and two weeks after, during a control visit, which is also associated with physical therapy. Thus, there are some discrepancies between the two procedures at the beginning of the treatment process.

It has been proven that intra- articular injection of autologous fat tissue or PRP is a safety treatment option of knee OA (49,50). The most common complications after the intra- articular injection are pain and swelling of treated knee, but this improve after cold compression and NSAIDs. Also there were no cancer incidents reported after autologous fat tissue or PRP implantation(50).

Subject recruitment has started after we received Bioethical Committee approval.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic knee OA
* Kellgren- Lawrence grades I - III OA
* no or minimal positive effects of previous conservative treatment (rehabilitation, hyaluronic acid injections, steroid injections)
* VAS pain level minimum 4 in one knee, VAS pain < 2 in the contralateral knee

Exclusion Criteria:

* Use of local corticosteroids up to three months or hyaluronic acid injections up to six months prior to the study
* Past or present joint infection
* Previous knee arthroscopy surgery up to one year prior to examination
* Peripheral inflammatory diseases (rheumatoid arthritis, spondyloarthropathies, etc.)
* Total arthroplasty and osteotomy
* Ankylosis of the joint
* Dermatitis or dermatological disease at the intended injection site
* Coexistence of degenerative changes in other limb joints (hip, foot)
* Cancer
* Oral corticosteroid therapy
* Use of medicines that affect blood clotting
* Pregnancy or breast-feeding

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in The Knee injury and Osteoarthritis Outcome Score (KOOS) | 1, 3, 6 and 12 months after the treatment
  The answers are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated.
Change in the International Knee Documentation Committee 2000 (IKDC 2000) score | 1, 3, 6 and 12 months after the treatment
  The IKDC contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Change in tthe Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score | 1, 3, 6 and 12 months after the treatment
  Due to no polish version of the WOMAC score, it will be calculated from KOOS score. Higher scores represent worse pain, stiffness, and functional limitations.
Change in the quality of life score (EQ- 5D- 5L) | 1, 3, 6 and 12 months after the treatment
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  Scores range from 5 points (highest level of function and lowest level of symptoms) to 25 points (lowest level of function or highest level of symptoms).
Change in functional status according to The Timed Up and Go Test (TUG) | 1, 3, 6 and 12 months after the treatment
  The result of this test is time measured with stopwatch. Time limit for this test is 3 minutes 30 seconds. Less time means better result.
Change in functional status according to The 5 Times Sit to Stand Test (5xSTS) | 1, 3, 6 and 12 months after the treatment
  The result of this test is time measured with stopwatch. The stopwatch is stopped when the subject sits down after the fifth repetition. Less time means better result.
Change in functional status according to The 10m Walk Test (10mWT) | 1, 3, 6 and 12 months after the treatment
  The result of this test is time measured with stopwatch. The patient is not allowed to run but may use the crutches or a walker if needed. Less time means better result.

SECONDARY OUTCOMES:
Strength parameters | 1, 3, 6 and 12 months after the treatment
  Strength parameters of the knee flexors and extensors the Maximal Voluntary Isometric Contraction (MVIC)

CONTACTS AND LOCATIONS:
Overall Officials: Pawel Bakowski, MD PhD, Principal Investigator — Rehasport Clinic; Tomasz Piontek, MD PhD, Study Chair — Rehasport Clinic
Locations (1):
- Rehasport, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bakowski P, Kaszynski J, Walecka J, Ciemniewska-Gorzela K, Bakowska-Zywicka K, Piontek T. Autologous adipose tissue injection versus platelet-rich plasma (PRP) injection in the treatment of knee osteoarthritis: a randomized, controlled study - study protocol. BMC Musculoskelet Disord. 2020 May 20;21(1):314. doi: 10.1186/s12891-020-03345-8. PMID 32434498